CLINICAL TRIAL: NCT06842810
Title: Evaluation of Serum Fibroblast Growth Factor 21 Levels in Patients With Systemic Lupus Erythematosus
Brief Title: Fibroblast Growth Factor 21 in Systemic Lupus Erythematosus
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Sayed Ibrahim Abdelrahman, Dr., Assiut University
Other Study IDs: Fibroblast growth factor 21
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Systemic Lupus Erthematosus
Keywords: SLE; Fibroblast growth factor 21

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- SLE cases with lupus nephritis
  Interventions: Diagnostic Test: Serum FGF21 measurement by Enzyme- linked immunosorbent assay (ELISA)
- SLE cases without lupus nephritis
  Interventions: Diagnostic Test: Serum FGF21 measurement by Enzyme- linked immunosorbent assay (ELISA)
- Healthy controls
  Interventions: Diagnostic Test: Serum FGF21 measurement by Enzyme- linked immunosorbent assay (ELISA)

INTERVENTIONS:
Diagnostic Test: Serum FGF21 measurement by Enzyme- linked immunosorbent assay (ELISA) — Venous 5 ml blood will be collected, then centrifugation at the speed of 2000-3000 rpm for 20-min., supernatant will be collected and stored at -20°C for later analysis then tha sample will be tested for fibroblast growth factor 21

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic disorder characterized by profound immune and metabolic disturbances. It emerges due to a complex interplay of genetic and environmental factors. Alteration in immune cell metabolism is another feature of SLE. Mitochondria, serving as the main regulator of cell metabolism, exhibits pronounced dysfunction in SLE patients.

Kidneys are among the most frequently affected organs in SLE, with 30-40% of patients developing lupus nephritis (LN) over the course of their disease. LN patients exhibit varying degrees of renal injury, significantly reducing their survival rate. Usually, LN originates from abnormal immune responses, resulting in the formation and deposition of immune complexes in the kidneys, triggering the release of pro-inflammatory cytokines, cell adhesion molecules, and chemokines, thereby inducing inflammation. Extensive glomerular mitochondrial damage has been reported in kidney biopsies obtained from patients with LN. So, identifying peripheral immune markers of mitochondrial dysfunction may be beneficial in assessing SLE activity and the extent of organ involvement.

Among these markers, fibroblast growth factor 21 (FGF-21) is one of the circulating immune markers which is expressed in response to mitochondrial stress. FGF-21 is known to be primarily produced in the liver, but under stress conditions, it can also be produced by the kidneys. In addition, it correlates with the degree of renal impairment in various kidney diseases.

ELIGIBILITY:
Inclusion Criteria:

- 1- Patients who will be diagnosed as SLE according to the 2019 EULAR/ACR Classification criteria for Systemic Lupus Erythematosus.

2-SLE Patients > 18 years old.

Exclusion Criteria:

* 1-SLE Patients < 18 years old. 2- Patients with other rheumatic diseases or overlap syndromes. 3- Patients with malignancy. 4- Patients with liver diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 50 SLE patients with lupus nephritis
  * 25 SLE patients without lupus nephritis
  * 20 healthy controls
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of serum FGF21 level in SLE patients with and without nephritis in comparison to healthy controls. | 2 years

IPD SHARING:
Plan to Share IPD: Undecided